CLINICAL TRIAL: NCT04072003
Title: Intravascular Ultrasound(IVUS) vs Angiography Guided Percutaneous Coronary Intervention(PCI) for Patients With Left Main Bifurcation Lesion
Brief Title: IVUS VS CAG Guided PCI for Patients With LMB Lesion
Acronym: Infinite
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Head of department of Cardiology, Zhongshan hospital, principal investigator, clinical professor, Shanghai Zhongshan Hospital
Other Study IDs: B2018246
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease; Left Main Coronary Artery Disease
Keywords: Left main, bifurcation, IVUS,PCI
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVUS-guided PCI: In this group, intravascular ultrasound(IVUS) in addition to coronary angiography(CAG) is used to guide percutaneous coronary intervention(PCI) procedure of left main bifurcation lesion.
  Interventions: Device: intravascular ultrasound (IVUS); Other: coronary angiography
- CAG-guided PCI: In this group, coronary angiography(CAG) is used to guide percutaneous coronary intervention(PCI) procedure of left main bifurcation lesion.
  Interventions: Other: coronary angiography

INTERVENTIONS:
Device: intravascular ultrasound (IVUS) — use IVUS in the procedure
  Groups: IVUS-guided PCI
Other: coronary angiography — Coronary angiography is required for all PCI procedure.

SUMMARY:
To compare the 3 - year clinical follow - up results of patients with left main bifurcation lesions treated by intravascular ultrasound(IVUS) - guided and coronary angiography(CAG) - guided percutaneous coronary intervention(PCI), and to confirm the clinical benefits of optimizing interventional therapy of left main bifurcation lesions by intravascular ultrasound(IVUS).

DETAILED DESCRIPTION:
616 patients with primary left main coronary artery bifurcation lesions will be recruited in this study. The target lesions of patients need to be true coronary artery bifurcation lesions (Medina 1,1,1 or 0,1,1). After angiography, patients will be randomly assigned to intravascular ultrasound(IVUS) - guided and coronary angiography (CAG)- guided groups. The random number of patients will be generated by the central computer random system, and the random will be stratified according to the study sites. In coronary angiography(CAG)-guided group, two-stent technique will be used(the exact two-stent technique used was left to the operator's discretion). In intravascular ultrasound(IVUS)-guided group, minimal lumen area(MLA) in ostium of side branch will be measured by intravascular ultrasound(IVUS). If minimal lumen area(MLA)<4mm2, two-stent technique will be used(the exact two-stent technique used was left to the operator's discretion) and intravascular ultrasound(IVUS) will be repeated at the end of the procedure. If minimal lumen area(MLA) >=4mm2, one-stent technique will be used and intravascular ultrasound(IVUS) will be repeated. If minimal lumen area(MLA) in ostium of side branch is still >=4mm2, the procedure will be ended. If minimal lumen area(MLA) in ostium of side branch become <4mm2, the following interventional strategy will be left to the operator's discretion( balloon inflation, drug-eluting balloon, or switch to two-stent technique). Again, intravascular ultrasound(IVUS) will be repeated at the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable or unstable angina pectoris, asymptomatic myocardial ischemia or attack of myocardial infarction >24 h;
2. True bifurcation lesion of left main coronary artery (Medina 1,1,1 or 0,1,1);
3. According to coronary angiography, the opening stenosis of the left anterior descending (LAD) and left circumflex (LCX) is more than 50% visually;
4. The operator judges that the lesion is suitable for drug eluting stent(DES) implantation;
5. Branch vessel diameter ≥2.5 mm by visual inspection;

Exclusion Criteria:

1. Pregnant or lactating women;
2. Combined with other diseases, life expectancy <1 year;
3. A surgery is scheduled within 6 months after the operation, and this surgery affects continuous administration of antiplatelet drugs;
4. The dual antiplatelet therapy cannot be tolerated;
5. Follow - up visits required by the protocol cannot be followed, or the investigators believe that the participation of subjects in the trial will increase the risk;
6. Unable to provide written informed consent form, or unable to follow the trial protocol;
7. Participate in another clinical trial of coronary interventional device;
8. Subjects with myocardial infarction within 24 h of onset of chest pain (including ST segment elevation or non - ST segment elevation);
9. Suffer from renal failure requiring dialysis treatment or is undergoing dialysis treatment;
10. Hemoglobin <9 g/L;
11. Uncontrolled hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥ 110 mmHg);
12. Severe cardiac insufficiency (LVEF <30%);
13. Heart failure complicated with pulmonary hypertension (mean pulmonary artery pressure(mPAP) ≥25 mmHg,pulmonary capillary wedge pressure (PCWP) >15 mmHg, and pulmonary vascular resistance (PVR)>3.0WU);
14. Complicated with hypertrophic obstructive cardiomyopathy;
15. Re-stenotic bifurcation lesion;
16. Severe calcified lesions requiring rotational atherectomy;
17. Chronic total occlusion lesion without successful recanalization;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary left main coronary artery bifurcation lesions will be recruited in this study. The target lesions of patients need to be true coronary artery bifurcation lesions (Medina 1,1,1 or 0,1,1)
Sampling Method: Probability Sample
Enrollment: 616 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure rate(the rate of outcomes including cardiac death, target vessel myocardial infarction(MI), and clinically driven main branch or side branch target vessel revascularization(TVR) in each group) | 12th month after stent implantation
  Cardiac death is defined as death resulting from an acute myocardial infarction (MI), sudden cardiac death, stroke, death due to heart failure (HF), death due to cardiovascular (CV) procedures, death due to CV hemorrhage, and death due to other CV causes; target vessel MI is defined as a MI case with the evidence of myocardial necrosis in the vascular territory of previously treated vessel; clinically driven main branch or side branch TVR is defined as a revascularization procedure with repeated stenting, balloon angioplasty or surgical bypass grafting for restenosed or occluded culprit target vessel.

SECONDARY OUTCOMES:
major adverse cardiac and cerebrovascular events（MACCE）rate（ the percentage of outcomes including all cause death, stroke, myocardial infarction(MI), and all clinically driven target vessel revascularization(TVR) in each group) | 30 days, 6 months, 12 months, 24 months and 36 months after operation
  TVR is defined as a revascularization procedure with repeated stenting, balloon angioplasty or surgical bypass grafting for restenosed or occluded culprit target vessel.
The percentage of in-stent restenosis (ISR) assessed by quantitative coronary angiography(QCA) in each group | 12 months after operation
  ISR is defined as a >50% stenosis of a previously stented segment as judged by QCA after coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No
Whether to share the data will be decided by the principal investigator